CLINICAL TRIAL: NCT00417924
Title: Eye Health and Vision Care for Patients With Diabetes: Comparing Usual Care to a Targeted Intervention in a Randomized Controlled Trial
Brief Title: Eye on Diabetes: A Multidisciplinary Patient Education Intervention
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: OPT06170409X
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2006-12

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Patient education; Patient satisfaction; Eye health
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Patient Satisfaction | interventions — Patient Education as Topic

INTERVENTIONS:
Behavioral: Patient education

SUMMARY:
Vision loss from diabetes is often preventable with timely detection and treatment. Patients with diabetes may not understand the importance of annual dilated eye examinations or recognize the benefits of early detection of diabetic eye disease. The proposed research project compares usual eye care to eye care emphasizing patient education for adult patients with diabetes.

DETAILED DESCRIPTION:
Patients with diabetes may not understand the importance of annual dilated eye examinations or recognize the benefits of early detection of diabetic eye disease. The goal of this study is to compare the efficacy of usual care to an intervention emphasizing patient education targeted at a multicultural adult patient population with diabetes seeking eye care in an academic health center. The specific aims of this study are to evaluate patient knowledge of preventive health strategies for diabetes as they pertain to eye health and vision care, to assess patient satisfaction with eye and vision care, and to promote interdisciplinary collaboration in the care of patients with diabetes.

Ninety patients were randomized to two arms representing usual care and an intervention emphasizing patient education targeted at English-speaking adults with diabetes seeking eye care in an academic health center. The project was developed within the Health Professions Division at Nova Southeastern University.

Participation was comprised of a comprehensive eye health and vision examination, patient education, and completion of study instruments described below. A demographic survey documenting patient age, sex, physician-reported HbA1C, education, and birthplace was administered to all patients at baseline. Race and ethnicity were self reported using categories in current use by the National Eye Institute, National Institutes of Health (Bethesda, MD).

Patients assigned to the intervention were provided with a written report at the conclusion of the examination. The triplicate form included a report of eye examination findings with a copy designated for the medical record, the primary care physician, and the patient. The back side of the patient's copy included educational materials targeted at a layperson while the physician's copy included information directed at a primary health care provider.

Patients assigned to usual care received patient education at the discretion of the eye care provider. Following the initial examination, all medical records were reviewed with attention to communication with other health care providers, as well as other issues related to continuity and coordination of care. Patients assigned to usual care were mailed additional written educational materials at the conclusion of the study, after all study instruments had been completed.

Patients assigned to the intervention were invited to participate in a supplementary seminar that reinforced the educational message delivered at the time of the initial examination. A multidisciplinary (optometry, pharmacy, endocrinology) patient education curriculum incorporating materials from the National Eye Health Education Program (NEHEP) Diabetic Eye Disease Public Education Program, the "ABC's of diabetes", an interactive activity, and a question and answer session was developed for patients randomized to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Type I or Type II Diabetes
* English speaking

Exclusion Criteria:

* Visual acuity worse than 20/60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-10; Study Completion 2005-10

PRIMARY OUTCOMES:
Patient knowledge (pre-test, post-test, and 3 month post-test)
Patient satisfaction post-examination

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Wagner, OD, MPH, Principal Investigator — Nova Southeastern University, Health Professions Division
Locations (1):
- Sanford L. Ziff Health Center, Fort Lauderdale, Florida, United States